CLINICAL TRIAL: NCT05671224
Title: Visual Aids for Induction of Labor (IOL): A Randomized Controlled Trial for Assessment of Patient IOL Knowledge
Brief Title: Visual Aids for Induction of Labor RCT
Acronym: VAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 202301001
Record Dates: First submitted 2023-01-01; First posted 2023-01-04 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Induced; Birth
MeSH Terms: interventions — Audiovisual Aids

STUDY DESIGN:
Intervention Model Description: Using a web-based randomization sequence on REDCap, patients will be randomized in 1:1 ratio to standard counseling or counseling with a visual aid immediately prior to initiation of their IOL.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard counseling (No Intervention): Standard induction of labor counseling
- Visual aid counseling (Experimental): Counseling on induction of labor with either a video or a handout
  Interventions: Other: Visual aid

INTERVENTIONS:
Other: Visual aid — Handout and video describing different types of induction of labor
  Arms: Visual aid counseling

SUMMARY:
This study aims to develop a visual aid tool for induction education informed by the experiences and needs of historically marginalized pregnant women, as well as determine the impact of the patient-informed visual aid on patient knowledge, satisfaction, and trust in physicians regarding induction methods.

DETAILED DESCRIPTION:
This is a multi-phased study of patients undergoing IOL. Only the second phase of the study will be detailed in this protocol, as this will be the RCT portion of the study's design. We will test the efficacy of the visual aid by conducting a randomized trial of routine counseling versus counseling with the use of a visual aid (informed by patient interviews in the first phase) at the time of admission for IOL and studying the effect of the visual aid on patient knowledge, trust in providers, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for or admitted for induction of labor and who can speak, read, and write in the English language.

Exclusion Criteria:

* Patients undergoing induction termination or with a history of prior cesarean section, major fetal anomaly, known chromosomal anomaly, or fetal growth restriction with doppler abnormalities. Patients whose induction has already commenced will also be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Induction of labor knowledge | 10 minutes (during completion of survey)
  Multiple choice questions

SECONDARY OUTCOMES:
Patient satisfaction | 10 minutes (during completion of survey)
  Likert scale (1-10)
Patient trust in providers survey | 10 minutes (during completion of survey)

CONTACTS AND LOCATIONS:
Overall Officials: Nandini Raghuraman, MD, MS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Beckmann M, Cooper C, Pocock D. INFORMed choices: facilitating shared decision-making in health care. Aust N Z J Obstet Gynaecol. 2015 Jun;55(3):294-7. doi: 10.1111/ajo.12343. Epub 2015 Jun 5. PMID 26053591
- [Background] Berger B, Schwarz C, Heusser P. Watchful waiting or induction of labour--a matter of informed choice: identification, analysis and critical appraisal of decision aids and patient information regarding care options for women with uncomplicated singleton late and post term pregnancies: a review. BMC Complement Altern Med. 2015 May 7;15:143. doi: 10.1186/s12906-015-0663-y. PMID 25947100
- [Background] Cahill AG, Tuuli MG, Stout MJ, Lopez JD, Macones GA. A prospective cohort study of fetal heart rate monitoring: deceleration area is predictive of fetal acidemia. Am J Obstet Gynecol. 2018 May;218(5):523.e1-523.e12. doi: 10.1016/j.ajog.2018.01.026. Epub 2018 Feb 1. PMID 29408586
- [Background] Irani RA, Foster S. Overview of the mechanisms of induction of labor. Semin Perinatol. 2015 Oct;39(6):426-9. doi: 10.1053/j.semperi.2015.07.001. Epub 2015 Sep 11. PMID 26372360
- [Background] Hamm RF, Srinivas SK, Levine LD. Risk factors and racial disparities related to low maternal birth satisfaction with labor induction: a prospective, cohort study. BMC Pregnancy Childbirth. 2019 Dec 30;19(1):530. doi: 10.1186/s12884-019-2658-z. PMID 31888529
- [Background] Bailey JM, Crane P, Nugent CE. Childbirth education and birth plans. Obstet Gynecol Clin North Am. 2008 Sep;35(3):497-509, ix. doi: 10.1016/j.ogc.2008.04.005. PMID 18760232
- [Background] Sperlich M, Gabriel C, St Vil NM. Preference, knowledge and utilization of midwives, childbirth education classes and doulas among U.S. black and white women: implications for pregnancy and childbirth outcomes. Soc Work Health Care. 2019 Nov-Dec;58(10):988-1001. doi: 10.1080/00981389.2019.1686679. Epub 2019 Nov 4. PMID 31682786
- [Background] Rosenthal L, Lobel M. Gendered racism and the sexual and reproductive health of Black and Latina Women. Ethn Health. 2020 Apr;25(3):367-392. doi: 10.1080/13557858.2018.1439896. Epub 2018 Feb 15. PMID 29447448
- [Background] Rahman S, Kripalani S, Keegan E, Sparks A, Amdur R, Moawad G, Sheth S, Klebanoff J. An educational video's impact on the induction of labor experience: a randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Jan;4(1):100495. doi: 10.1016/j.ajogmf.2021.100495. Epub 2021 Sep 24. PMID 34571210
- [Background] Anderson LA, Dedrick RF. Development of the Trust in Physician scale: a measure to assess interpersonal trust in patient-physician relationships. Psychol Rep. 1990 Dec;67(3 Pt 2):1091-100. doi: 10.2466/pr0.1990.67.3f.1091. PMID 2084735